CLINICAL TRIAL: NCT03833973
Title: The Evaluation of Cell-Free Plasma DNA (cfDNA) and Oxidative Stress Indices as Biomarkers for the Diagnosis and Prevention of Overtraining
Brief Title: Safety and Prevention of OveRTraining
Acronym: SuPpOrt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Other Study IDs: SuPpOrt-UTH
Record Dates: First submitted 2018-06-05; First posted 2019-02-07 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Overtraining Syndrome
Keywords: Training; Cell free plasma DNA; Oxidative stress; Performance
MeSH Terms: conditions — Overtraining Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Runners: Long-distance runners, marathon runners, 5 km and 10 km runners, both female and male aged 20 - 40 years, participating in regular training and competitions.
  Interventions: Behavioral: Overtraining Monitoring
- Soccer Players: High Level soccer players, both female and male aged 15-30, participating in all games
  Interventions: Behavioral: Overtraining Monitoring

INTERVENTIONS:
Behavioral: Overtraining Monitoring — Athletes will be thoroughly monitored (i.e. training workload, match activities or event/race performance, markers of inflammation and oxidative stress as well as cell-free DNA) throughout the season in order to establish novel biomarkers that could function as either predictors or diagnostic tools of overtraining.

SUMMARY:
Athletic training aims to increase and improve physical performance that is achieved through training overload combined with periods of rest and recovery. Overtraining syndrome (OTS) is associated with an imbalance between training and recovery. The symptoms associated with OTS vary between individuals and may reflect parasympathetic and/or sympathetic nervous system alterations as well as endocrine irregularities. The prevalence is not known, but it is usually reported among endurance athletes, such as cyclists, distance runners and triathletes. It appears that OTS represents a systemic inflammatory process with diffuse effects on the neurohormonal axis affecting host immunology and mood. Previous works, showed that cell-free DNA (cf-DNA) is correlated with the severity of excessive exercise-induced inflammation as well as with trauma and stroke severity suggesting that it might be used as a potential clinical marker for athletes with overtraining syndrome. Oxidative stress indices can be determined non-invasively and may reflect inflammatory responses after training suggesting that they could be used as clinical markers for the diagnosis of OTS. However, there are no available biomarkers to aid towards the diagnosis and/or prevention of OTS, except that of the persistence of unexplained underperformance despite an extensive recovery of the athlete. Therefore, the purpose of this study is to evaluate the potential of cf-DNA and selected oxidative stress variables as diagnostic biomarkers of OTS.

DETAILED DESCRIPTION:
A total number of 15 elite-level runners (both male and female) and 80-100 soccer players (both male and female) will participate in the study.The day when participants (runners) will arrive at the lab early in the morning, after an overnight fast. They will have their blood pressure and orthostatic heart rate measured and they will also provide a blood sample. Immediately after participants' body composition will be assessed by dual energy X-ray absorptiometry (DXA). Then, they will perform the Meeusen test providing a second blood sample immediately after the test. During the subsequent 4-hour resting period, the participants followed by assessment of joint mobility, delayed onset of muscle soreness, flexibility and vertical jump performance after that lower limb peak torque by isokinetic dynamometer. A second Meeusen test will take place after the resting period with blood sampling post-testing. Then, participants will have a 3-hour rest, after which they will visit the lab again in order to perform the running economy testing protocol and a maximal lactate steady state test. Finally, participants will complete POMS-, quality of sleep- and symptomatology-related questionnaires and will be taught on how to complete dietary recalls. Over the subsequent 12-month period participants will provide the investigator with a detailed report of their training plan and a symptomatology questionnaire every month. These measurements take place for all participants in two different periods, in transitional period/baseline and in middle season (berore tha main race). If someone of participants manifest the symptoms of overtraining, they perform the protocol of measurements again. The day when participants (soccer players) will arrive at the lab early in the morning, after an overnight fast. They will have their blood pressure and orthostatic heart rate measured and they will also provide a blood sample. Immediately after participants' body composition will be assessed by dual energy X-ray absorptiometry (DXA). The participants followed by assessment of joint mobility, delayed onset of muscle soreness, flexibility and vertical jump performance after that lower limb peak torque by isokinetic dynamometer. After resting, they will measurement the maximum oxygen uptake in stress test on the aisle. The next days, in football players take place in field tests, will measure the Speed in 10, 30 meters, Yo-Yo IE2 (Intermittent Endurance 2), Yo-Yo IR2 (Intermittent Recovery 2) and Repeated Sprint Ability (RSA). Finally, participants (soccer players) will complete POMS-, quality of sleep- and symptomatology-related questionnaires and will be taught on how to complete dietary recalls.These measurements take place for all participants in two different periods, in transitional period/baseline and in middle season (berore tha main race). If someone of participants manifest the symptoms of overtraining, they perform the protocol again.

ELIGIBILITY:
Inclusion Criteria for Runners:

Participants:

* should be long-distance runners, marathon runners, 5 km and 10 km runners.
* should be able to provide the daily training plan and a 7-day dietary recall every month.
* should be considered elite level runners.
* should be free of musculoskeletal injuries for at least one year before the study.

Inclusion Criteria for Soccer Players:

Participants:

* should be elite soccer players.
* should be able to provide the daily training plan and a 7-day dietary recall.
* should be participated in matches.
* should be free of musculoskeletal injuries for at least one year before the study.

Exclusion Criteria (both Runners and Soccer Players):

If participants:

* do not adhere to rules of the study.
* have a recent history of illness or injury .
* do not participate in competitive training.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants for the first group will be male and female long-distance, marathon, 5 km and 10 km runners aged 20-40 years. All of them will be active, elite-level runners , participating in regular competitive training. For the second group will be male and female high level soccer players aged 15-30 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in cell free plasma DNA | At baseline, at six months and at twelve months
  Cell free plasma DNA will be measured with real-time PCR in plasma samples.
Change in Cortisol level | At baseline, at six months and at twelve months
  Cortisol concentration will measured in serum
Change in Testosterone level | At baseline, at six months and at twelve months
  Testosterone concentration will be measured in serum
Change in cytokine response | At baseline, at six months and at twelve months
  Concentration of TNF-α, IL-6 and IL-10 will be measured in plasma.
Change in creatine kinase in plasma | At baseline, at six months and at twelve months
  Concentration of creatine kinase will be measured in plasma
Change in uric acid in plasma | At baseline, at six months and at twelve months
  Concentration of uric acid will be measured in plasma
Change in protein carbonyls in blood | At baseline, at six months and at twelve months
  Concentration of protein carbonyls will be measured in red blood cells
Change in total antioxidant capacity | At baseline, at six months and at twelve months
  Total antioxidant capacity will be measured in plasma
Change in reduced glutathione in blood | At baseline, at six months and at twelve months
  Concentration of reduced glutathione will be measured in in red blood cells
Change in oxidized glutathione in blood | At baseline, at six months and at twelve months
  Concentration of oxidized glutathione will be measured in red blood cells
Change in catalase activity | At baseline, at six months and at twelve months
  Catalase activity will be measured in red blood cells
Change in malondialdehyde in blood | At baseline, at six months and at twelve months
  Concentration of malondialdehyde will be measured in serum

SECONDARY OUTCOMES:
Change in blood lactate concentration | At baseline, at six months and at twelve months
  Blood lactate concentration will be measured during a maximal lactate steady-state test.
Change in peak torque | At baseline, at six months and at twelve months
  Peak torque will be assessed on an isokinetic dynamometer at 60 degrees/sec
Change in orthostatic heart rate. | At baseline, at six months and at twelve months
  Heart rate will be measured in a resting position and following 15 seconds of standing by heart rate monitor.
Change in jumping ability. | At baseline, at six months and at twelve months
  Jumping ability will be assessed by measuring squat jump.
Change in flexibility | At baseline, at six months and at twelve months
  Flexibility will be assessed through the sit and reach test.
Change in body composition. | At baseline, at six months and at twelve months
  Body composition will be assessed by dual energy X-ray absorptiometry (DXA)
Change in delay onset of muscle soreness (DOMS) | At baseline, at six months and at twelve months
  DOMS will be assessed by muscle palpation while participants are laying , standing and after performing 3 squats.
Change in complete blood count | At baseline, at six months and at twelve months
  Complete blood count analysis will be performed on an automatic blood analyzer.
Change in RSA | At baseline, at six months and at twelve months
  5 x 30 m sprints will be performed with 25 seconds rest in-between. Mean time for 5 sprints and fatigue index will be calculated.
Change in Yo-Yo IE2 | At baseline, at six months and at twelve months
  Yo-Yo IE2 will be assessed using a standardized testing protocol.
Change in Yo-Yo IR2 | At baseline, at six months and at twelve months
  Yo-Yo IR2 will be assessed using a standardized testing protocol.
Change in Spreed | At baseline, at six months and at twelve months
  Spreed will be assessed using a standardized testing protocol in 10 and 30 meters.
Dietary intake | At baseline, at six months and at twelve months
  Dietary intake will be assessed using 7-day diet recalls.
Change in jumping ability. | At baseline, at six months and at twelve months
  Jumping ability will be assessed by measuring counter-movement jump.
Change in jumping ability. | At baseline, at six months and at twelve months
  Jumping ability will be assessed by measuring drop jump.

CONTACTS AND LOCATIONS:
Overall Officials: Vasiliki C Laschou, PhDc, Principal Investigator — UNIVERSITY OF THESSALY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Trikala, Greece